CLINICAL TRIAL: NCT01983566
Title: Investigation of the Effect of Food and of Increased Gastric pH on the Relative Bioavailability of Deleobuvir Following Single Oral Administration in Healthy Caucasian and Japanese Subjects (an Open-label, Randomised, Four-way Crossover Study)
Brief Title: Effect of Food and Increased Gastric pH Value on Bioavailability of a Single Dose of BI 207127 in Healthy Caucasian and Japanese Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1241.44; 2013-003967-74 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-11-05; First posted 2013-11-14 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — deleobuvir; Omeprazole

ARMS (4):
- BI 207127 fasted (Active Comparator): patient to receive BI 207127 as a single dose in fasted state
  Interventions: Drug: BI 207127
- BI 207127 high fat (Experimental): patient to receive BI 207127 as a single dose after a high fat breakfast
  Interventions: Drug: BI 207127 high fat
- BI 207127 low fat (Experimental): patient to receive BI 207127 as a single dose after a low fat breakfast
  Interventions: Drug: BI 207127 low fat
- BI 207127 with Omeprazole (Experimental): patient to receive BI 207127 as a single dose after 4 days treatment with Omeprazole 40 mg once a day
  Interventions: Drug: BI 207127 with Omeprazole

INTERVENTIONS:
Drug: BI 207127 high fat — BI 207127 as a single dose after a high fat breakfast
  Arms: BI 207127 high fat
Drug: BI 207127 with Omeprazole — BI 207127 as a single dose after 4 days treatment of Omeprazole 40 mg once a day
  Arms: BI 207127 with Omeprazole
Drug: BI 207127 — BI 207127 as a single dose in fasted state
  Arms: BI 207127 fasted
Drug: BI 207127 low fat — BI 207127 as a single dose after a low fat breakfast
  Arms: BI 207127 low fat

SUMMARY:
The purpose of this trial is to investigate the effect of food with different fat content and of gastric pH increase (mediated by multiple dosing of omeprazole) on the relative bioavailability of deleobuvir.

ELIGIBILITY:
Inclusion criteria:

* Healthy males or females according to the investigators assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests. Subjects will be either Caucasian or Japanese (first generation Japanese: born in Japan with parents of Japanese descent, and not more than 5 years out of Japan, documented by medical interview and by appropriate materials - e.g. passport, birth certificate, etc)
* Age 20 to 35 years (incl.)
* BMI 18.5 to 25 kg/m2 (incl.)

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
* Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
* Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.44.49001 Boehringer Ingelheim Investigational Site, Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned that 16 healthy Caucasian subjects (males and females, at least one third of each sex) and 16 healthy Japanese subjects (both males + females, at least one third of each sex) would enter the study. They were recruited from the volunteers' pool of the trial site. Due to early study termination, no Japanese subjects were randomised.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that the subject met all strictly implemented inclusion/exclusion criteria.
  Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat: Each subject received a single dose of 3 x 200 mg Deleobuvir (Dele) film-coated tablets after an overnight fast of at least 10 hours (h), followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised high-fat, high-calorie meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h after 4 days of pre-treatment with a 40 mg Omeprazole (OMP) gastro-resistant hard capsule once daily, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised low-fat meal after an overnight fast of at least 10 h.
  All medications were administered oral with 240 mL of water.
- Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised high-fat, high-calorie meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised low-fat meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h after 4 days of pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily.
  All medications were administered oral with 240 mL of water.
- Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised low-fat meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h after 4 days of pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised high-fat, high-calorie meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h.
  All medications were administered oral with 240 mL of water.
- Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h after 4 days of pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised low-fat meal after an overnight fast of at least 10 h, followed by a washout phase of at least 6 days; then each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised high-fat, high-calorie meal after an overnight fast of at least 10 h.
  All medications were administered oral with 240 mL of water.
Period: Test Period 1
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Wash-Out 1
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Test Period 2
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Wash-Out 2
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 2 (Subjects starting may not equal number completing the previous period due to early study termination) | 3 (Subjects starting may not equal number completing the previous period due to early study termination) | 2 (Subjects starting may not equal number completing the previous period due to early study termination) | 4
Completed | 2 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Test Period 3
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 2 | 3 | 2 | 4
Completed | 2 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Wash-Out 3
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 0 (Subjects starting may not equal number completing the previous period due to early study termination) | 0 (Subjects starting may not equal number completing the previous period due to early study termination) | 0 (Subjects starting may not equal number completing the previous period due to early study termination) | 0 (Subjects starting may not equal number completing the previous period due to early study termination)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Test Period 4
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): included all subjects who were dispensed study medication and were documented to have taken at least 1 dose of deleobuvir or OMP.
Groups:
- Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat: Dele fasted, followed by a washout phase, followed by Dele after a standardised high-fat, high- calorie meal, followed by a washout phase, followed by Dele after a 4 days pre-treatment with a 40 mg Omeprazole (OMP) gastro-resistant hard capsule once daily, followed by a washout phase, followed by Dele after a standardised low-fat meal.
  Each Dele intake is a single dose of 3x 200mg Dele film-coated tablets after an overnight fast of at least 10 h.
  The duration of a washout phase was at least 6 days.
- Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP: Dele after a standardised high-fat, high-calorie meal, followed by a washout phase, followed by Dele after a standardised low-fat meal, followed by a washout phase, followed by Dele fasted, followed by a washout phase, followed by Dele after a 4 days pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily.
  Each Dele intake is a single dose of 3x 200mg Dele film-coated tablets after an overnight fast of at least 10 h.
  The duration of a washout phase was at least 6 days.
- Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted: Dele after a standardised low-fat meal, followed by a washout phase, followed by Dele after a 4 days pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily, followed by a washout phase, followed by Dele after a standardised high-fat, high-calorie meal, followed by a washout phase, followed by Dele fasted.
  Each Dele intake is a single dose of 3x 200mg Dele film-coated tablets after an overnight fast of at least 10 h.
  The duration of a washout phase was at least 6 days.
- Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat: Dele after a 4 days pre-treatment with a 40 mg OMP gastro-resistant hard capsule once daily, followed by a washout phase, followed by Dele fasted, followed by a washout phase, followed by Dele after a standardised low-fat meal, followed by a washout phase, followed by Dele after a standardised high-fat, high-calorie meal.
  Each Dele intake is a single dose of 3x 200mg Dele film-coated tablets after an overnight fast of at least 10 h.
  The duration of a washout phase was at least 6 days.
- Total: Total of all reporting groups
Arm/Group | Dele Fasted / Dele High Fat / Dele + OMP / Dele Low Fat | Dele High Fat / Dele Low Fat / Dele Fasted / Dele + OMP | Dele Low Fat / Dele + OMP / Dele High Fat / Dele Fasted | Dele + OMP / Dele Fasted / Dele Low Fat / Dele High Fat | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (3.0) | 25.3 (1.0) | 32.3 (2.9) | 27.8 (3.0) | 28.6 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 0 | 7
  Male | 2 | 2 | 1 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tz)
Description: Area under the concentration-time curve of deleobuvir in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz)
Time Frame: 1 hour (h) before drug administration and 30 minutes (min), 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h and 48h after drug administration
Population: Pharmacokinetic set (PKS): included all subjects in the Treated Set who provided at least 1 observation for at least 1 primary pharmacokinetic (PK) endpoint that was not affected by important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Dele Fasted: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h.
  The tablets were administered oral with 240 mL of water.
- Dele High Fat: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised high-fat, high-calorie meal after an overnight fast of at least 10 h.
  The tablets were administered oral with 240 mL of water.
- Dele Low Fat: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after a standardised low-fat meal after an overnight fast of at least 10 h.
  The tablets were administered oral with 240 mL of water.
- Dele + OMP: Each subject received a single dose of 3 x 200 mg Dele film-coated tablets after an overnight fast of at least 10 h after 4 days of pre-treatment with a 40 mg Omeprazole (OMP) gastro-resistant hard capsule once daily.
  All medications were administered oral with 240 mL of water.
Arm/Group | Dele Fasted | Dele High Fat | Dele Low Fat | Dele + OMP
Number analyzed (Participants) | 11 | 10 | 12 | 10
nmol*h/L | 9790 (60.2) | 16900 (98.8) | 14200 (46.8) | 15800 (72.1)
Statistical Analysis 1: Comparison: Dele Fasted vs Dele Low Fat; The difference between the expected means for log(Dele low fat) and log(Dele fasted) was estimated by the differences in the adjusted means (Least Squares Means), and a 2 sided 90% confidence interval (CI) based on the t-distribution was computed. These were then back transformed. The estimation model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'; Test type: Non-Inferiority or Equivalence — The actual number of subjects analyzed is 16. No formal statistical hypothesis was tested; p = 0.3944, ANOVA — The p-value relates to the null hypothesis of non-equivalence (bioequivalence test). P-value for ratio outside interval 80-125%; Geometric mean ratio (%) = 115.80, 90% CI 2-sided [63.52 to 211.11] — This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'. The statistical analysis result is based on the adjusted means

2. Primary Outcome: Cmax
Description: Maximum measured concentration of deleobuvir in plasma (Cmax)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Dele Fasted | Dele High Fat | Dele Low Fat | Dele + OMP
Number analyzed (Participants) | 11 | 10 | 12 | 10
nmol/L | 2140 (60.1) | 3930 (92.5) | 3160 (52.2) | 3190 (90.2)
Statistical Analysis 1: Comparison: Dele Fasted vs Dele Low Fat; The difference between the expected means for log(Dele low fat) and log(Dele fasted) was estimated by the differences in the adjusted means (Least Squares Means), and a 2 sided 90% CI based on the t-distribution was computed. These were then back transformed. This estimation model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'; Test type: Non-Inferiority or Equivalence — The actual number of subjects analyzed is 16. No formal statistical hypothesis was tested; p = 0.3674, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio (%) = 114.83, 90% CI 2-sided [74.803 to 176.281] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC(0-inf)
Description: Area under the concentration-time curve of deleobuvir in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf)
Time Frame: as for outcome 1
Population: PKS - Due to premature discontinuation of the study, this endpoint was not evaluated.
Arm/Group | Dele Fasted | Dele High Fat | Dele Low Fat | Dele + OMP
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of first administration of the respective treatment until start of the next treatment or until the day after the termination date (or until 3 days after administration of last study drug, whichever occurred later), up to 37 days.
Groups:
- OMP Alone: One gastro-resistant hard capsule of Omeprazole (OMP) (40 mg) once daily in the evening for 4 days administered oral with 240 mL of water.
Arm/Group | Dele Fasted | Dele High Fat | Dele Low Fat | Dele + OMP | OMP Alone
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/11 | 1/10 | 4/12 | 7/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dele Fasted (N=11) | Dele High Fat (N=10) | Dele Low Fat (N=12) | Dele + OMP (N=10) | OMP Alone (N=10)
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
As the study was discontinued prematurely, the results were incomplete. Due to this incomplete data the endpoint AUC(0-inf) was not evaluated,and only a limited number of the planned statistical analyses could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.